CLINICAL TRIAL: NCT02790294
Title: Optimal Timing of Postoperative Magnetic Resonance Imaging (MRI) in Patients With Extradural Spinal Tumors - a Pilot Study
Brief Title: Optimal Timing of Postoperative Magnetic Resonance Imaging (MRI) in Patients With Extradural Spinal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE4314
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Spinal Tumor
Keywords: magnetic resonance imaging
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postoperative Magnetic Resonance Imaging (Experimental): Three MRIs will be performed. One at baseline, one within 72 hours postoperative, and one 2-3 weeks postoperative.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — The routine spine MRI protocol will be utilized, which includes the following sequences: haste localizer, sagittal T1, T2, and short-T1 Inversion Recovery (STIR), axial T2 for lumbar spine or axial gradient echo for cervical and thoracic spine, axial T1, post contrast sagittal and axial T1. All scans will be obtained using a 1.5 Tesla magnet.
  Other Names: MRI

SUMMARY:
This research study is evaluating suitability of a delayed magnetic resonance imaging (MRI) in management of spine tumors. Currently the standard of care is obtaining an MRI scan in the early postoperative period (within 72 hours after surgery). The purpose of this study is to see if delayed MRI (2 to 3 weeks after surgery) is similar in quality to the earlier MRI.

In this study patients will undergo 2 MRIs after the surgery instead of one MRI. Patients will have one MRI about 3 days after the surgery and one MRI about 2-3 weeks after surgery.

DETAILED DESCRIPTION:
Primary aim:

Assess if Magnetic Resonance Imaging (MRI) at 2 to 3 weeks after surgery leads to the same clinical decisions and has the same probability of being chosen by a physician for guiding the subsequent management of the patient, compared with immediately postoperative MRI.

Secondary aims:

Investigate the differences between early and late MRI by comparing:

* Size of tumor in three dimensions;
* Extent of edema;
* Presence and extent of fluid collection;
* Spine Oncology Study Group score;
* Involvement of adjacent levels;
* Progression of tumor;
* Patient's preference/performance scale right after each image had taken: level of discomfort at around the time each MRI was performed.

Study Design:

This is a prospective diagnostic study for which no standard of care currently exists.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or primary malignant tumor involving spinal column, with or without extension into the epidural space
* Operated for debulking, decompression or separation surgery;
* A magnetic resonance imaging (MRI) scan performed within 72 hours after surgery is needed;
* Image quality acceptable for comparison with later MRI as read by a neuroradiologist;
* Karnofsky score of 60 or higher;
* Able to consent for the study.

Exclusion Criteria:

* Any patient who previously underwent spinal surgery at these levels will be excluded to eliminate late postoperative changes.
* Intradural extension of the tumor.
* Patients, whose MRI at post operative 48-72 hours are not readable due to artifacts or disease process shall not be included in the study.
* Patient not able to tolerate MRI scan due to claustrophobia or severe pain or allergic reaction to contrast.
* Patients with an estimated Glomerular Filtration Rate (eGFR) < or = to 30 will be excluded to avoid issues related to contrast administration in such patients. This Glomerular Filtration Rate (GFR) threshold cutoff level is chosen per institutional policy, because below that level other measures would be required (hydration or no contrast administration). In order to keep the imaging information as uniform as possible in such a small study group, patients with a low GFR will not be enrolled in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Number of patients which have the same clinical decision from the immediate postoperative MRI and later imaging | Up to 3 weeks after surgery
  Assess if Magnetic Resonance Imaging (MRI) at 2 to 3 weeks after surgery (aka: later imaging) leads to the same clinical decisions and has the same probability of being chosen by a physician for guiding the subsequent management of the patient, compared with immediately postoperative MRI (within 72 hours, aka: early imaging).

SECONDARY OUTCOMES:
Change in tumor volume between immediate and later postoperative MRI | Up to 3 weeks after surgery
Difference in level of discomfort as measured by a visual analog scale between postoperative MRIs | Up to 3 weeks after surgery
Progression of tumor using RECIST Criteria | Up to 3 weeks after surgery
  RECIST response categories: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.

CONTACTS AND LOCATIONS:
Overall Officials: Lilyana Angelov, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States